CLINICAL TRIAL: NCT01456195
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Daily Oral TAK-875 25 mg and 50 mg Compared With Placebo in Subjects With Type 2 Diabetes
Brief Title: Comparison of TAK-875 (Fasiglifam) With Placebo in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_301; 2011-002741-35 (EudraCT Number); U1111-1124-2154 (Registry Identifier: WHO)
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Fasiglifam placebo-matching tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: Placebo
- Fasiglifam 25 mg (Experimental): Fasiglifam 25 mg, tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: Fasiglifam
- Fasiglifam 50 mg (Experimental): Fasiglifam 50 mg, tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: Fasiglifam

INTERVENTIONS:
Drug: Placebo — Fasiglifam placebo-matching tablets
  Arms: Placebo
Drug: Fasiglifam — Fasiglifam tablets
  Arms: Fasiglifam 25 mg; Fasiglifam 50 mg

SUMMARY:
The purpose of this study is to determine the efficacy and safety of TAK-875 (fasiglifam), once daily (QD), in participants with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
TAK-875 is being developed at Takeda Development Center, Inc. as an adjunct to diet and exercise to improve glycemic control in patients with T2DM.

This study will investigate TAK-875 in participants with type 2 diabetes mellitus who have been treated with only diet and exercise for at least 12 weeks prior to Screening, who have taken ≤7 days of any antidiabetic agent within the 12 weeks prior to Screening, and whose glycemic control is inadequate.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is male or female and 18 years of age or older with a historical diagnosis of T2DM.
4. The participant has been treated with only diet and exercise for at least 12 weeks prior to Screening and has an HbA1c concentration between 7.0 % and 10.5%, inclusive, at Screening.
5. The participant has received ≤7 days of any antidiabetic agent within 12 weeks prior to Screening.
6. The participant has a body mass index (BMI) ≤45 kg/m^2 at Screening.
7. Participants regularly using other, non-excluded medications must be on a stable dose for at least 4 weeks prior to Screening. However, as needed (PRN) use of prescription or over-the-counter medication is allowed at the discretion of the investigator.
8. The participant is able and willing to monitor glucose with a home glucose monitor and consistently record his or her own blood glucose concentrations and complete participant diaries.
9. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of the informed consent throughout the duration of the study and for 30 days after the last dose of study drug.

Additional Inclusion Criteria prior to Randomization

1. The participant has an HbA1c concentration between 7.0 and 10.5%, inclusive, and a fasting plasma glucose (FPG) ≤270 mg/dL (≤15.0 mmol/L) at Week -1 Visit. (If the participant does not qualify for randomization based on these criteria, the assessments may be repeated weekly, for a maximum of 2 additional weeks).
2. The participant's overall compliance with single-blind study medication during the Placebo Run-in Period is at least 75% and does not exceed 125% based on tablet counts performed by the study staff.
3. A female participant of childbearing potential must have a negative urine hCG pregnancy test at Baseline (Visit 4) prior to Randomization and prior to administration of the first dose of double-blind study medication

Exclusion Criteria:

1. The participant has received any investigational compound within 30 days prior to Screening or has received an investigational antidiabetic drug within 3 months prior to Screening.
2. The participant has been randomized in a previous TAK-875 study.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, or sibling; biological or legally adopted) or may consent under duress.
4. The participant donated or received any blood products within 12 weeks prior to Screening or is planning to donate blood during the study.
5. The participant has a hemoglobin ≤12 g/dL (≤120 gm/L) for males and ≤10 g/dL (≤100 gm/L) for females at Screening.
6. The participant has a systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥95 mm Hg at Screening (If the participant meets this exclusion criterion, the assessment may be repeated once at least 30 minutes after the initial measurement and decision will be made based on the second measurement).
7. The participant has a history of cancer that has been in remission for <5 years prior to Screening. A history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed.
8. The participant has an alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >2.0x the upper limit of normal (ULN) at Screening.
9. The participant has a total bilirubin level greater than the ULN at Screening. Exception: if a participant has documented Gilbert's Syndrome, the participant will be allowed with an elevated bilirubin level per the investigator's discretion.
10. The participant has a serum creatinine ≥1.5 mg/dL(≥133 µmol/L) [males] and ≥1.4 mg/dL (≥124 µmol/L) [females] and/or estimated glomerular filtration rate (GFR) <60 mL/min/1.73m^2 at Screening.
11. The participant has uncontrolled thyroid disease.
12. The participant has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
13. The participant has had gastric banding or gastric bypass surgery within one year prior to Screening.
14. The participant has a known history of infection with human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
15. The participant had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram (ECG), cerebrovascular accident or transient ischemic attack within 3 months prior or at Screening.
16. The participant has a history of hypersensitivity, allergies, or has had an anaphylactic reaction(s) to any component of TAK-875.
17. The participant has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse within 2 years prior to Screening.
18. The participant received excluded medications prior to Screening or is expected to receive excluded medication.
19. If female, the participant is pregnant (confirmed by laboratory testing, i.e., serum human chorionic gonadotropin (hCG), in females of childbearing potential) or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
20. The participant is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.
21. The participant has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the participant according to the protocol.

Additional Exclusion Criteria prior to Randomization

1. The participant received excluded medications during the Placebo Run-in Period. (Topical and inhaled corticosteroids are allowed).
2. The participant has a systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥95 mm Hg at Baseline (Visit 4) (If the participant meets this exclusion criterion, the assessment may be repeated once at least 30 minutes after the initial measurement and decision will be made based on the second measurement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Takeda
Locations (95):
- United States (55):
  - Dothan, Alabama
  - Muscle Shoals, Alabama
  - Goodyear, Arizona
  - Phoenix, Arizona
  - Long Beach, California
  - North Hollywood, California
  - Norwalk, California
  - Palm Springs, California
  - Pismo Beach, California
  - Boynton Beach, Florida
  - Bradenton, Florida
  - Coral Gables, Florida
  - Hialeah, Florida
  - Largo, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Avon, Indiana
  - Greenfield, Indiana
  - Muncie, Indiana
  - Council Bluffs, Iowa
  - Topeka, Kansas
  - Lexington, Kentucky
  - Oxon Hill, Maryland
  - Flint, Michigan
  - Picayune, Mississippi
  - Omaha, Nebraska
  - Elizabeth, New Jersey
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Mooresville, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Maumee, Ohio
  - Oklahoma City, Oklahoma
  - Harleysville, Pennsylvania
  - Levittown, Pennsylvania
  - Uniontown, Pennsylvania
  - Greer, South Carolina
  - Crossville, Tennessee
  - Carrollton, Texas
  - Dallas, Texas
  - El Pasco, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Manassas, Virginia
- Argentina (6):
  - Buenos Aires, Ciudad Autonoma Buenos Aires
  - Ciudad Autonoma Buenos Aires, Ciudad Autonoma Buenos Aires
  - Corrientes, Corrientes Province
  - Córdoba, Córdoba Province
  - Villa Cabrera, Córdoba Province
  - Mendoza, Mendoza Province
- Bulgaria (5):
  - Byala
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Guatemala (3):
  - Guatemala City
  - Quetzaltenango
  - Zacapa
- Hungary (6):
  - Budapest
  - Debrecen
  - Kecskemét
  - Komárom
  - Szikszó
  - Zalaegerszeg
- Mexico (2):
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
- Slovakia (10):
  - Banská Bystrica
  - Bratislava
  - Dolný Kubín
  - Komárno
  - Levice
  - Pezinok
  - Prievidza
  - Trebišov
  - Trenčín
  - Žilina
- Ukraine (8):
  - Dnipropetrovsk
  - Kharkiv
  - Kyiv
  - Odesa
  - Simferopol
  - Ternopil
  - Vinnytsia
  - Zaporizhzhia

REFERENCES:
- [Derived] Shavadia JS, Sharma A, Gu X, Neaton J, DeLeve L, Holmes D, Home P, Eckel RH, Watkins PB, Granger CB. Determination of fasiglifam-induced liver toxicity: Insights from the data monitoring committee of the fasiglifam clinical trials program. Clin Trials. 2019 Jun;16(3):253-262. doi: 10.1177/1740774519836766. Epub 2019 Mar 18. PMID 30880443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 109 investigative sites in United States, Bulgaria, Argentina, Ukraine, Guatemala, Slovakia, Mexico and Hungary from 02 November 2011 to 30 July 2013.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitis were enrolled equally in 1 of 3 treatment groups, once a day placebo, 25 mg fasiglifam or 50 mg fasiglifam.
Period: Overall Study
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Started | 143 | 137 | 141
Completed | 132 | 127 | 127
Not Completed | 11 | 10 | 14
Not completed — Pretreatment Event/Adverse Event | 1 | 4 | 1
Not completed — Lost to Follow-up | 3 | 1 | 3
Not completed — Voluntary Withdrawal | 5 | 3 | 7
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Other Reasons | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg | Total
Number analyzed (Participants) | 143 | 137 | 141 | 421
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.61) | 53.2 (11.31) | 54.2 (10.57) | 53.5 (10.82)
Age, Customized [Number; unit: participants]
  < 65 years | 124 | 114 | 114 | 352
  ≥ 65 years | 19 | 23 | 27 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 65 | 73 | 206
  Male | 75 | 72 | 68 | 215
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 22 | 25 | 22 | 69
  Non-Hispanic or Latino | 39 | 36 | 41 | 116
  Not Applicable | 82 | 76 | 78 | 236
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 19 | 15 | 16 | 50
  Asian | 5 | 4 | 0 | 9
  Black or African American | 8 | 6 | 12 | 26
  White | 110 | 112 | 113 | 335
  Multiracial | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Argentina | 10 | 10 | 10 | 30
  Bulgaria | 8 | 7 | 9 | 24
  Guatemala | 15 | 14 | 13 | 42
  Hungary | 8 | 7 | 8 | 23
  Mexico | 6 | 5 | 7 | 18
  Slovakia | 24 | 24 | 24 | 72
  Ukraine | 11 | 9 | 8 | 28
  United States | 61 | 61 | 62 | 184
Height [Mean (Standard Deviation); unit: cm] | 166.3 (10.63) | 165.3 (11.17) | 166.7 (11.11) | 166.1 (10.96)
Weight [Mean (Standard Deviation); unit: kg] | 89.66 (18.858) | 89.24 (18.541) | 89.43 (18.706) | 89.45 (18.660)
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.33 (5.714) | 32.50 (5.256) | 32.05 (5.369) | 32.29 (5.443)
Baseline BMI Group [Number; unit: participants]
  < 30 kg/m^2 | 54 | 49 | 56 | 159
  ≥ 30 kg/m^2 | 89 | 88 | 85 | 262
Baseline HbA1c Category [Number; unit: participants]
  < 8.5% | 102 | 91 | 102 | 295
  ≥ 8.5 % | 41 | 46 | 39 | 126
Smoking Classification [Number; unit: participants]
  Never smoked | 99 | 98 | 97 | 294
  Current smoker | 21 | 17 | 23 | 61
  Ex-smoker | 23 | 22 | 21 | 66
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 3.048 (3.164) | 3.290 (3.447) | 3.700 (4.560) | 3.345 (3.773)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 24 relative to Baseline. A mixed model repeated measures (MMRM) model with treatment, country, visit and visit by treatment interaction as fixed factors and with Baseline value and Baseline value by visit interaction as covariates with an unstructured covariance structure was used for analysis.
Time Frame: Baseline and Week 24
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug, with data available for analysis. Only participants with Baseline and at least 1 post-Baseline value are included.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 101 | 119 | 116
percent | -0.17 (0.090) | -0.65 (0.087) | -0.93 (0.087)
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — MMRM model with treatment, country, visit and visit by treatment interaction as fixed factors and with baseline value and baseline value by visit interaction as covariates with an unstructured covariance structure; LS Mean Difference = -0.48, 95% CI 2-sided [-0.72 to -0.24], Standard Error of Mean 0.122
Statistical Analysis 2: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.76, 95% CI 2-sided [-1.00 to -0.52], Standard Error of Mean 0.122

2. Secondary Outcome: Incidence of HbA1c <7%
Description: The incidence (percentage of participants with) HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) of less than seven percent for target glycemic control at Week 24.
Time Frame: Week 24
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug, with data available for analysis. Only participants with Baseline and at least 1 post-Baseline value are included. Last Observation Carried Forward.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 137 | 136 | 139
percentage of participants | 24.1 | 36.0 | 50.4
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p = 0.010, Regression, Logistic — P-Value used a logistic model with treatment, country and baseline HbA1c as explanatory variables; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.20 to 3.79]
Statistical Analysis 2: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-Value used a logistic model with treatment, country and baseline HbA1c as explanatory variables; Odds Ratio (OR) = 4.40, 95% CI 2-sided [2.48 to 7.82]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change between the fasting plasma glucose value collected at Week 24 relative to Baseline measured in milligrams per deciliter (mg/dL). A MMRM model with treatment, country, visit and visit by treatment interaction as fixed factors and with Baseline value and Baseline value by visit interaction as covariates with an unstructured covariance structure was used for analysis.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 101 | 116 | 116
mg/dL | 1.4 (3.45) | -12.3 (3.29) | -20.9 (3.26)
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p = 0.003, Mixed model for repeated measurements — Mixed Model Repeated Measures (MMRM) model with treatment, country, visit and visit by treatment interaction as fixed factors and with baseline value and baseline value by visit interaction as covariates with an unstructured covariance structure; LS Mean Difference = -13.7, 95% CI 2-sided [-22.7 to -4.6], Standard Error of Mean 4.59
Statistical Analysis 2: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -22.3, 95% CI 2-sided [-31.4 to -13.2], Standard Error of Mean 4.60

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Glucose (PPG) Following a Meal Tolerance Test (MTT)
Description: The change between the value of glucose after a meal, measured by the meal tolerance test collected at Week 24 relative to Baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and 2 hours after the start of the meal measured in millimoles per liter (mmol/L). An Analysis of Covariance (ANCOVA) model with treatment and country as fixed factors and Baseline value as covariate was used for analysis.
Time Frame: Baseline and Week 24
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug, with data available for analysis. Only participants with Baseline and at least 1 post-Baseline value are included. MTT were only done at sites that had MTT capabilities.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 18 | 20 | 18
mmol/L | -0.6 (12.47) | -29.4 (11.82) | -30.6 (12.50)
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p = 0.100, ANCOVA — ANCOVA model with treatment and country as fixed factors and baseline value as covariate; LS Mean Difference = -28.8, 95% CI 2-sided [-63.2 to 5.7], Standard Error of Mean 17.17
Statistical Analysis 2: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p = 0.096, ANCOVA — ANCOVA model with treatment and country as fixed factors and baseline value as covariate; LS Mean Difference = -30.0, 95% CI 2-sided [-65.5 to 5.5], Standard Error of Mean 17.70

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days past last dose of study drug (Up to 28 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Fasiglifam 25 mg | Fasiglifam 50 mg
Serious Adverse Events (participants affected / at risk) | 3/143 | 3/137 | 3/141
Other Adverse Events (participants affected / at risk) | 9/143 | 6/137 | 7/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=143) | Fasiglifam 25 mg (N=137) | Fasiglifam 50 mg (N=141)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=143) | Fasiglifam 25 mg (N=137) | Fasiglifam 50 mg (N=141)
Nasopharyngitis (Infections and infestations) | 9 | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.